CLINICAL TRIAL: NCT01462929
Title: A Multiple Dose, Double-blind, Double-dummy, Placebo Controlled, Parallel Clinical Trial to Assess the Efficacy and Safety of Twice Daily Inhaled Aclidinium Bromide 400 µg Compared to Placebo and to Tiotropium Bromide in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Aclidinium Bromide 400 µg Compared to Placebo and to Tiotropium Bromide in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/39
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; antimuscarinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aclidinium bromide (Experimental): Aclidinium bromide 400 µg administered twice per day during 6 weeks of treatment
  Interventions: Drug: Aclidinium bromide
- Tiotropium (Active Comparator): Tiotropium bromide 18 µg administered once per day during 6 weeks of treatment
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator): Placebo comparator administered during 6 weeks of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide — Dosage form: Dry powder. Route of administration: Oral inhalation by Genuair multidose dry powder inhaler Dose and regimen: 1 puff of 400 micrograms in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h)
  Arms: Aclidinium bromide
Drug: Tiotropium — Dosage form: Dry powder hard gelatin capsule. Route of administration: Oral inhalation by HandiHaler single-dose dry powder inhaler Dose and regimen: 1 capsule (18 μg) in the morning (09:00 ± 1h)
  Arms: Tiotropium
Drug: Placebo — Dosage form: Dry powder Route of administration: Oral inhalation by Genuair multidose dry powder inhaler. 1 puff of placebo in the morning (09:00 ± 1h) and 1 puff in the evening (21:00 ± 1h) AND Oral inhalation by HandiHaler single-dose dry powder inhaler. 1 puff of placebo in the morning (09:00 ± 1h).
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the 24h bronchodilatory efficacy of inhaled aclidinium bromide 400 µg administered twice a day versus placebo and tiotropium bromide, respectively, after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients aged ≥40 with stable moderate to severe COPD (GOLD guidelines).
* Post-salbutamol (FEV1) < 80% and ≥ 30% of predicted normal value and Post-salbutamol FEV1/FVC < 70%.
* Current or ex-smokers of 10 ≥pack-years.

Exclusion Criteria:

* Patients with no history or current diagnosis of asthma.
* No evidence of an exacerbation within 6 weeks prior to the screening visit.
* No evidence of clinically significant respiratory and/or cardiovascular conditions or laboratory abnormalities.
* No contraindication to use of anticholinergic drugs such as known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, Ph.D., Study Director — AstraZeneca
Locations (41):
- Czechia (3):
  - Almirall Investigational Site #9, Humpolec
  - Almirall Investigational Site #1, Jaroměř
  - Almirall Investigational Site #3, Mělník
- Germany (20):
  - Almirall Investigational Site #4, Berlin
  - Almirall Investigational Site #12, Berlin
  - Almirall Investigational Site #10, Berlin
  - Almirall Investigational Site #8, Berlin
  - Almirall Investigational Site #20, Berlin
  - Almirall Investigational Site #21, Berlin
  - Almirall Investigational Site #2, Berlin
  - Almirall Investigational Site #24, Cologne
  - Almirall Investigational Site #13, Dresden
  - Almirall Investigational Site #9, Frankfurt
  - Almirall Investigational Site #3, Großhansdorf
  - Almirall Investigational Site #1, Hamburg
  - Almirall Investigational Site #18, Hamburg
  - Almirall Investigational Site #5, Hanover
  - Almirall Investigational Site #22, Hanover
  - Almirall Investigational Site #14, Jena
  - Almirall Investigational Site #17, Lübeck
  - Almirall Investigational Site #23, Rüdersdorf
  - Almirall Investigational Site #6, Schwerin
  - Almirall Investigational Site #16, Wiesbaden
- Hungary (5):
  - Almirall Investigational Site #4, Debrecen
  - Almirall Investigational Site #2, Komárom
  - Almirall Investigational Site #3, Mátraháza
  - Almirall Investigational Site #1, Szarvas
  - Almirall Investigational Site #11, Szigetszentmiklós
- Poland (13):
  - Almirall Investigational Site #18, Bialystok
  - Almirall Investigational Site #8, Bialystok
  - Almirall Investigational Site #2, Elblag
  - Almirall Investigational Site #17, Krakow
  - Almirall Investigational Site #10, Krakow
  - Almirall Investigational Site #16, Lodz
  - Almirall Investigational Site #20, Lodz
  - Almirall Investigational Site #4, Proszowice
  - Almirall Investigational Site #6, Sopot
  - Almirall Investigational Site #14, Tarnów
  - Almirall Investigational Site #19, Warsaw
  - Almirall Investigational Site #12, Wilkowice-Bystra
  - Almirall Investigational Site #13, Wroclaw

REFERENCES:
- [Derived] McGarvey L, Morice AH, Smith JA, Birring SS, Chuecos F, Seoane B, Jarreta D. Effect of aclidinium bromide on cough and sputum symptoms in moderate-to-severe COPD in three phase III trials. BMJ Open Respir Res. 2016 Dec 8;3(1):e000148. doi: 10.1136/bmjresp-2016-000148. eCollection 2016. PMID 28074135
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3975&filename=Synopsis-las39-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 49 sites investigators in 4 countries (3 sites in the Czech Republic, 23 in Germany, 8 in Hungary and 15 in Poland). 8 sites (3 in Germany, 3 in Hungary and 2 in Poland) did not randomise any patients. The first patient was screened in Oct 2011 and the last patient visit was in Mar 2012.
Pre-assignment Details: Patients fulfilling inclusion/exclusion criteria at the time of the screening visit were entered into a run-in period of 14-21 days to assess disease stability.
Groups:
- Aclidinium Bromide 400 µg BID: Aclidinium bromide 400 µg administered twice per day
  Dosage form: Dry powder. Route of administration: Oral inhalation by Genuair multidose dry powder inhaler.
  Dose and regimen: 1 puff of 400 micrograms in the morning (09:00 ± 1h) and in the evening (21:00 ± 1h)
  AND
  1 capsule of placebo in the morning (09:00 ± 1h) via oral inhalation by HandiHaler single-dose dry powder inhaler.
- Tiotropium 18 μg Once-daily: Tiotropium 18 μg administered once daily
  Dosage form: Dry powder hard gelatin capsule. Route of administration: Oral inhalation by HandiHaler single-dose dry powder inhaler.
  Dose and regimen: 1 capsule (18 μg) in the morning (09:00 ± 1h)
  AND
  1 puff of placebo in the morning (09:00 ± 1h) and 1 puff in the evening (21:00 ± 1h) via oral inhalation by Genuair multidose dry powder inhaler.
- Placebo: Placebo
  Route of administration:
  Oral inhalation by Genuair multidose dry powder inhaler. 1 puff of placebo in the morning (09:00 ± 1h) and 1 puff in the evening (21:00 ± 1h) AND Oral inhalation by HandiHaler single-dose dry powder inhaler. 1 capsule of placebo in the morning (09:00 ± 1h).
Period: Overall Study
Arm/Group | Aclidinium Bromide 400 µg BID | Tiotropium 18 μg Once-daily | Placebo
Started | 171 | 158 | 85
Completed | 166 | 154 | 80
Not Completed | 5 | 4 | 5
Not completed — Adverse Event | 3 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 400 µg BID | Tiotropium 18 μg Once-daily | Placebo | Total
Number analyzed (Participants) | 171 | 158 | 85 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.2) | 62.8 (7.9) | 62.2 (8.2) | 62.3 (8.1)
Gender [Count of Participants; unit: Participants]
  Female | 57 | 42 | 37 | 136
  Male | 114 | 116 | 48 | 278
Region of Enrollment [Number; unit: participants]
  Hungary | 18 | 16 | 10 | 44
  Czech Republic | 5 | 3 | 3 | 11
  Poland | 64 | 58 | 32 | 154
  Germany | 84 | 81 | 40 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalised Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve Over the 24-h Period After 6 Weeks of Treatment
Description: Change from baseline in normalised FEV1 area under the curve over the 24-h period immediately after morning Investigational Medicinal Product administration (AUC0-24h ) after 6 weeks on treatment. The normalised AUC were calculated by means of a trapezoidal method, dividing by the corresponding time interval.
Time Frame: Week 6
Population: Intention to treat (ITT) population: patients who took at least 1 dose of Investigational Medicinal Product and had at least a baseline FEV1 assessment and at least one post-baseline FEV1 value
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 400 µg BID | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 170 | 158 | 85
Liters | 0.065 (0.017) | 0.055 (0.018) | -0.085 (0.023)

2. Secondary Outcome: Change From Baseline in Normalised FEV1 Area Under the Curve Over the 12-h Night-time Period After 6 Weeks of Treatment
Description: Change from baseline in normalised FEV1 area under the curve over the 12-h night-time period (AUC12-24) after 6 weeks of treatment. The normalised AUC were calculated by means of a trapezoidal method, dividing by the corresponding time interval.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 400 µg BID | Tiotropium 18 μg Once-daily | Placebo
Number analyzed (Participants) | 170 | 158 | 85
Liters | 0.032 (0.017) | -0.006 (0.018) | -0.128 (0.024)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: A follow-up was performed by means of a visit or a phone contact, as considered appropriate, 2 weeks (±3 days) after the last Investigational Medicinal Product dose administration in order to assess new or ongoing AEs, abnormal values of study variables (laboratory evaluations, BP or ECG) or COPD exacerbation.
Arm/Group | Aclidinium Bromide 400 µg BID | Tiotropium 18 μg Once-daily | Placebo
Serious Adverse Events (participants affected / at risk) | 3/171 | 4/158 | 0/85
Other Adverse Events (participants affected / at risk) | 16/171 | 17/158 | 6/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 400 µg BID (N=171) | Tiotropium 18 μg Once-daily (N=158) | Placebo (N=85)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Per protocol, only COPD exacerbations (worsening of COPD symptoms for at least 2 consecutive days that required a change in the patient's COPD treatment) were reported as AEs
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 400 µg BID (N=171) | Tiotropium 18 μg Once-daily (N=158) | Placebo (N=85)
Nasopharyngitis (Infections and infestations) | 11 | 8 | 2
Headache (Nervous system disorders) | 6 | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.